CLINICAL TRIAL: NCT05675709
Title: Enhancing Skin Cancer Early Detection and Treatment in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan A. Flocke, Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00024809; NCI-2022-09484 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00024809 (Other: OHSU Knight Cancer Institute); P50CA244289 (NIH)
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group (No Intervention): PCPs at the two clinics who do not receive the group training will serve as study comparators.
- Other, Pragmatic (Experimental): PCP participants complete group training. All training participants will also be offered series of short booster teaching points delivered virtually. Participants who complete the training also take part in pre-post knowledge assessments. PCP participants may also participate in a qualitative interview.
  Interventions: Behavioral: Training and Education

INTERVENTIONS:
Behavioral: Training and Education — Undergo group trainings
  Arms: Other, Pragmatic

SUMMARY:
Skin cancer screening may help find melanoma sooner, when it may be easier to treat. If found early melanoma and other types of skin cancer may be curable. Multi-component education may be an effective method to help primary care physicians (PCPs) learn about skin cancer screening. This clinical trial examines whether a clinician-focused educational intervention can improve PCP's knowledge and clinical performance to identify and triage skin cancer. This intervention may increase the PCP's ability to diagnose, treat and/or triage early-stage melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate whether a multi-component education strategy improves the ability of PCPs to identify and triage skin cancer.

OUTLINE:

Participants are assigned to 1 of 2 groups.

PCP participants complete group training. All training participants will also be offered series of short booster teaching points delivered virtually. Participants who complete the training also take part in pre-post knowledge assessments. PCP participants may also participate in a qualitative interview.

PCPs at the two clinics who do not receive the group training will serve as study comparators.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians at two Oregon Health & Science University (OHSU) primary care clinics will be invited to receive exposure to the melanoma early detection intervention
* Clinicians at the two clinics who do not receive the intervention will serve as study comparators
* These individuals are all aged 18 years or older
* All practice members speak English

Exclusion Criteria:

* No one will be intentionally excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Flocke, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No plan is needed

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five clinicians (physicians, PAs, and NPs) received an email inviting them to participate in the MelaNOma training. Seventeen participated in the training. A total of 37 clinicians who weren't invited or chose not to participate in the MelaNOma training session were assigned to the comparator group. The total study sample size is 54.
Groups:
- Melanoma Training Group: MelaNOma included a 40-minute hybrid training co-led by a family medicine physician and a dermatologist
- Comparison Group: Clinicians from the same 2 clinics who weren't invited or chose not to participate in the MelaNOma training session
Period: Overall Study
Arm/Group | Melanoma Training Group | Comparison Group
Started | 17 | 37
Completed | 15 | 29
Not Completed | 2 | 8
Not completed — incomplete outcome data | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Training Group: PCP participants complete group training. All training participants will also be offered series of short booster teaching points delivered virtually. Participants who complete the training also take part in pre-post knowledge assessments. PCP participants may also participate in a qualitative interview.
  Training and Education: Undergo group trainings
- Total: Total of all reporting groups
Arm/Group | Comparison Group | Training Group | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 15 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 11 | 5 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Knowledge in Melanoma Risk and Lesion Identification
Description: KnChange in melanoma risk, knowledge based upon survey questions prior to training and post-training. Content covered melanoma risk, knowledge of electronic health record tools specific to the training and lesion identification and biopsy procedure knowledge. A total score of correct responses for the 27 items was generated and transformed to represent the percent of correct items with zero being no correct items and 100% being all items correct. A change score from pre-training to post-training was generated where a positive change score represented the gain in knowledge in percent points and a negative change score representing a lower percent of correct responses from pre-training to post-training.
Time Frame: Immediately before and after the training session
Population: Knowledge was assessed before and after the training session for those clinicians who attended the training. We conducted a paired t-test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comparison group | Training group
Number analyzed (Participants) | 0 | 10
score on a scale
  Immediately before the training |  | 72.1 (7.2)
  Immediately after the training |  | 80.8 (9.6)
Statistical Analysis 1: Comparison: Training group; Test type: Superiority — paired t-test; p = 0.05, paired t-test

2. Primary Outcome: Dermatology Referral
Description: Mean percent of dermatology referrals per 1000 patients
Time Frame: minimum of 3 months and up to 1 year of EHR data for each clinician prior to the start of the training and the same months in the year post-training.
Measure: Mean (Standard Deviation); unit: percent per 1000 patients
Arm/Group | Comparison group | Training group
Number analyzed (Participants) | 29 | 15
percent per 1000 patients
  pre-training period | 13.8 (9.2) | 16.9 (9.0)
  post-training period | 14.1 (11.1) | 11.4 (6.7)
Statistical Analysis 1: Comparison: Comparison group vs Training group; Test type: Superiority; p = .05, generalized estimating equation (GEE)

3. Primary Outcome: Use of Dermatology E-consults
Description: number of dermatology e-consults
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent per 1000 patients
Arm/Group | Comparison group | Training group
Number analyzed (Participants) | 29 | 15
percent per 1000 patients
  pre-training period | 5.1 (7.8) | 5.5 (7.8)
  post-training period | 7.2 (9.2) | 7.8 (7.5)
Statistical Analysis 1: Comparison: Comparison group vs Training group; Test type: Superiority; p = .05, generalized estimating equation (GEE)

ADVERSE EVENTS:
Time Frame: Adverse event data from exposure to the training module was collected over 12 months.
Description: Adverse events to participating in the educational training module was assessed using a post training survey and during qualitative interviews with the 11 clinicians who agreed to participate in a debriefing interview.
Arm/Group | Comparison group | Training group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/17
Other Adverse Events (participants affected / at risk) | 0/29 | 0/17

LIMITATIONS AND CAVEATS:
The initial plan to randomize pods of clinicians within each of the two clinics proved not to be feasible and participation in the training module was much lower than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT05675709/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT05675709/SAP_001.pdf